CLINICAL TRIAL: NCT06546787
Title: The Effect of Interpersonal Relationships Psychotherapy on Depression, Emotion Regulation and Social Support Levels in Breast Cancer Patients With Depression Risk: A Randomized Controlled Study
Brief Title: The Effect of Interpersonal Relationships Psychotherapy on Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0036315
Record Dates: First submitted 2024-02-23; First posted 2024-08-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Patients Diagnosed
Keywords: Depression; Emotion Regulation; Social Support; Interpersonal Relationships; Breast Cancer
MeSH Terms: conditions — Depression; Emotional Regulation; Breast Neoplasms | interventions — Psychotherapy; Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychotherapy (Experimental): IPT will be administered by the researcher who has completed the interpersonal relations psychotherapy training.
  Interventions: Other: PSYCHOTHERAPY
- Observation (No Intervention): Patients in the control group will be asked to complete the post-tests at the same time after the experimental group interviews are completed. However, no intervention will be made to the control group.

INTERVENTIONS:
Other: PSYCHOTHERAPY — IPT, was prepared by the researcher who completed the interpersonal relations psychotherapy training.The first interview will be conducted face-to-face in the offices of Koç University Faculty of Nursing. Subsequent sessions will be conducted via Zoom according to the availability of the patients included in the study. The day and time of the interviews will be planned according to the availability of the patients before the interviews. A total of 12 interviews are planned to be conducted with a patient for 40-60 minutes each. Interview intervals will be organized as once a week.
  Other Names: interpersonal psychotherapy
  Arms: Psychotherapy

SUMMARY:
This study is planned to examine the effect of Interpersonal Relationship Psychotherapy on depression, interpersonal emotion regulation and multidimensional perceived social support levels of breast cancer patients with depression risk.

DETAILED DESCRIPTION:
There are not enough studies showing the effect of IPT, which is an evidence-based psychotherapy that works on problem areas such as role change that may occur with the disease and provides support for recognizing and using social support mechanisms, on cancer patients. This study is thought to make a significant contribution to the literature, especially in terms of making family support, which has an important place in social support systems, available to patients, intervening in interpersonal emotion regulation problems that may occur in patients and affecting depression levels.

ELIGIBILITY:
Includes Criteria

* Ability to communicate in Turkish
* Diagnosed with Stage-II and Stage-III breast cancer
* Continuing outpatient treatment
* Four points on the Primary Care Depression Screening Scale
* Internet connection
* Has a phone that can use the zoom app to continue conversations to be
* To be able to use the Zoom app

Exclusion Criteria

* Being a pediatric oncology/hematology patient
* Diagnosed with stage -IV breast cancer
* Taking psychopharmacological medication
* To have received KIPT within the last year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Screening Scale for Primary Care | Through study completion, an average of 6 months
  Each question has four answers. The lowest possible score is zero and the highest possible score is three. A total maximum score of 21 and a minimum score of zero can be achieved. Depression scores of breast cancer patients are expected to decrease after treatment. It is expected to fall below 4 points.
Interpersonal relationships emotion regulation scale | Through study completion, an average of 6 months
  The highest score that can be obtained from the scale is 100 and the lowest score is 20. The high score obtained from each sub-dimension of the scale indicates that the individual has the characteristic evaluated by the relevant sub-dimension. Scores obtained from the scale were found to be related to the total score of the Difficulties in Emotion Regulation Scale and also to depression and anxiety.An increase in the interpersonal relations emotion regulation scale score is expected in breast cancer patients after treatment. This increase shows that it has a positive effect on individuals' emotion regulation.
Multidimensional Perceived Social Support Scale: | Through study completion, an average of 6 months
  The lowest score that can be obtained from the scale is "12" and the highest score is "84". An increase in the total score of the scale means an increase in the level of perceived social support. Social support scores of breast cancer patients are expected to increase after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University, Istanbul, Nursing Department, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No